CLINICAL TRIAL: NCT02715037
Title: Mikrobiologi Ved svær Akut Tonsillit, peritonsillær Phlegmone og infektiøs Mononukleose
Brief Title: Microbiology of Severe Acute Tonsillitis, Peritonsillar Cellulitis, and Infectious Mononucleosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tejs Ehlers Klug (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor-Investigator, Tejs Ehlers Klug, Consultant, associate professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: 52683
Record Dates: First submitted 2016-03-14; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Acute Tonsillitis; Peritonsillar Cellulitis; Infectious Mononucleosis
Keywords: fusobacterium necrophorum; acute tonsillitis; peritonsillar cellulitis; infectious mononucleosis; microbiology; antibody development
MeSH Terms: conditions — Infectious Mononucleosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Throat swabs Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Acute tonsillitis: Patients referred to the tertiary care center with severe acute tonsillitis but without peritonsillar cellulitis, infectious mononucleosis, or abscess formation.
  Interventions: Other: Throat swabbing
- Peritonsillar cellulitis: Patients referred to the tertiary care center with severe acute tonsillitis and peritonsillar cellulitis but without abscess formation.
  Interventions: Other: Throat swabbing
- Infectious mononucleosis: Patients referred to the tertiary care center with acute tonsillitis and biochemical or serological signs of infectious mononucleosis but without abscess formation.
  Interventions: Other: Throat swabbing
- Controls: Patients treated for conditions not related to the throat and without signs or symptoms of recent throat disease.
  Interventions: Other: Throat swabbing

INTERVENTIONS:
Other: Throat swabbing
  Other Names: Blood sample

SUMMARY:
Prospective, observational study of the microbiology of patients referred to a tertiary care center with severe acute tonsillitis, peritonsillar cellulitis, or infectious mononucleosis.

DETAILED DESCRIPTION:
Patients referred to tertiary care centers with acute throat infections are most often treated with antibiotics. However, very little is know concerning the prevalent pathogens in patients with acute throat infections without abscess formation. Evidence suggests that Fusobacterium necrophorum plays an important role in complications of acute tonsillitis (e.g. peritonsillar abscess), but also uncomplicated acute tonsillitis.

This study aims to explore the throat microbiology of patients with severe acute tonsillitis, peritonsillar cellulitis, or infectious mononucleosis with a special attention to a possible role of Fusobacterium necrophorum.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to our tertiary care center with acute tonsillitis with or without signs of peritonsillar cellulitis and with or without infectious mononucleosis.
2. Center Score 3 or 4.

Exclusion Criteria:

1. Abscess formation.
2. Previous tonsillectomy.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 100 patients with severe acute tonsillitis 100 patients with peritonsillar cellulitis 50 patients with infectious mononucleosis
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Fusobacterium necrophorum in throat swab cultures | At acute consultation (day 0)

SECONDARY OUTCOMES:
Number of participants with recurrent throat infections (questionnaire) | Six months after acute consultation
Number of participants without eradication of throat pathogens (throat cultures) | 14-28 days after acute consultation
  "Throat pathogens": Fusobacterium necrophorum, Beta-hemolytical streptococci, A. hemolyticum
Number of participants with complications of severe acute tonsillitis, peritonsillar cellulitis, and infectious mononucleosis | 14-28 days after acute consultation
  "Complications": admission, abscess Development, change of antibiotic treatment
Prevalence of anti-Fusobacterium necrophorum antibody Development (two-fold or higher increase in antibody level) (blood samples) | In acute and convalescent sera (day 0 and 14-28)
  Comparison of the prevalence of antibody Development (two-fold or higher increase in antibody level) between patients with recovery of Fusobacterium necrophorum in throat swabs versus patients without recovery of Fusobacterium necrophorum in throat swabs

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klug TE, Henriksen JJ, Rusan M, Fuursted K, Krogfelt KA, Ovesen T, Struve C. Antibody development to Fusobacterium necrophorum in patients with peritonsillar abscess. Eur J Clin Microbiol Infect Dis. 2014 Oct;33(10):1733-9. doi: 10.1007/s10096-014-2130-y. Epub 2014 May 9. PMID 24810966
- [Background] Klug TE. Incidence and microbiology of peritonsillar abscess: the influence of season, age, and gender. Eur J Clin Microbiol Infect Dis. 2014 Jul;33(7):1163-7. doi: 10.1007/s10096-014-2052-8. Epub 2014 Jan 29. PMID 24474247
- [Background] Klug TE, Henriksen JJ, Fuursted K, Ovesen T. Significant pathogens in peritonsillar abscesses. Eur J Clin Microbiol Infect Dis. 2011 May;30(5):619-27. doi: 10.1007/s10096-010-1130-9. Epub 2010 Dec 22. PMID 21181222
- [Background] Ehlers Klug T, Rusan M, Fuursted K, Ovesen T. Fusobacterium necrophorum: most prevalent pathogen in peritonsillar abscess in Denmark. Clin Infect Dis. 2009 Nov 15;49(10):1467-72. doi: 10.1086/644616. PMID 19842975